CLINICAL TRIAL: NCT01884727
Title: A Randomized, Cross-Over Clinical Trial to Evaluate the Acute Effects of ASEA on Energy Expenditure and Fat Oxidation in Humans
Brief Title: Effect of ASEA on Energy Expenditure and Fat Oxidation in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12-1675
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Over nutrition; nutrition disorders; energy expenditure; metabolic rate
MeSH Terms: conditions — Obesity; Overweight; Nutrition Disorders | interventions — Fluoridation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASEA water (Active Comparator): Subjects to consume 4-ounces of ASEA water at 9:00 am before breakfast and 4-ounces of ASEA water at 10:15 pm prior to bedtime. 24-h resting energy expenditure and RQ to be measured.
  Interventions: Dietary Supplement: ASEA water
- Salt water (Placebo Comparator): Subjects to consume 4-ounces of salt water at 9:00 am before breakfast and 4-ounces of salt water at 10:15 pm prior to bedtime. 24-h resting energy expenditure and RQ to be measured.
  Interventions: Dietary Supplement: Salt Water

INTERVENTIONS:
Dietary Supplement: Salt Water — Subjects to arrive fasted and will spend two 24-h periods inside the metabolic chamber (ASEA or salt water) with a one week interval between visits. Blood will be drawn at 9 am prior to consumption of salt water or breakfast, and at 11 am after consumption of salt water and breakfast. Subjects will receive a second portion of salt water at 10:15 pm just prior to bedtime. The energy content of meals will be identical at each visit.
  Arms: Salt water
Dietary Supplement: ASEA water — Subjects to arrive fasted and will spend two 24-h periods inside the metabolic chamber (ASEA or salt water) with a one week interval between visits. Blood will be drawn at 9 am prior to consumption of ASEA water or breakfast, and at 11 am after consumption of ASEA water and breakfast. Subjects will receive a second portion of ASEA water at 10:15 pm just prior to bedtime. The energy content of meals will be identical at each visit.
  Arms: ASEA water

SUMMARY:
To test the effect of ASEA consumption on 24-hour resting energy expenditure. Hypothesis: consumption of 8-oz of ASEA water (4-oz before breakfast and 4-oz before bedtime) will significantly elevate 24-h resting energy expenditure as compared to consumption of a placebo control (salt water, same dietary intake).

DETAILED DESCRIPTION:
The ASEA beverage is a special oral formulation produced from a pure saline solution containing 123 mg sodium and 129 mg chloride per 4 oz. serving. A proprietary electrolytic and catalytic process rearranges the salt water solution to mimic the redox signaling molecular composition of the native salt-water compounds found in and around human cells. Data obtained thus far, suggests the possibility that consumption of the ASEA beverage may increase energy expenditure and thus be beneficial for the treatment of obesity, however, this has not been assessed in human clinical studies. To this end, we will measure the effects of ASEA consumption on energy expenditure by indirect calorimetry using the indirect room calorimeter at the University of North Carolina (UNC) Nutrition Research Institute.

The primary outcome measures will be the change in 24-h energy expenditure and respiratory quotient in response to ASEA consumption. The secondary outcome variables will include changes in relevant peptide hormones, and norepinephrine/epinephrine and their relationship to changes in energy expenditure in response to consumption of ASEA.

ELIGIBILITY:
Inclusion Criteria:

* woman
* postmenopausal
* healthy
* age 50-65
* BMI 25-35 kg/m²
* exercise less than 150 minutes per week
* weight neutral for past 6 months

Exclusion Criteria:

* smoker
* exercises more than 150 minutes per week
* abuses drugs or alcohol
* vegetarian
* taking herbal supplements, attention deficit hyperactivity disorder (ADHD) medication or thyroid medication
* taking beta-blockers, steroidal anti-inflammatory medication
* taking pseudoephedrine

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure | 24-hours
  Changes in 24-h resting energy expenditure and respiratory quotient (RQ) in response to ASEA or control salt water to be measured by indirect calorimetry in the room indirect calorimeter at the UNC Nutrition Research Institute.

SECONDARY OUTCOMES:
Plasma Hormones | 0900 and 1100 hours
  Relevant peptide hormones and nor-epinephrine/epinephrine will be assessed before consumption of ASEA (or control water) before breakfast (9:00 am) and after consumption of ASEA (or control water) after breakfast (11:00 am).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Swick, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Nutrition Research Institute, Kannapolis, North Carolina, United States